CLINICAL TRIAL: NCT03628365
Title: Can Beta-Hydroxy-beta-Methylbutyrate (HMB) Supplementation Counteract Muscle Catabolism in Critically Ill Patients? A Randomized Controlled Trial
Brief Title: Can Beta-Hydroxy-beta-Methylbutyrate Supplementation Counteract Muscle Catabolism in Critically Ill Patients?
Acronym: HMB-ICU-CH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mette M Berger (Other)
Collaborators: Texas A&M University (Other)
Responsible Party: Sponsor-Investigator, Mette M Berger, Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CER-2018-00556
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Critical Illness; Muscle Weakness
Keywords: Body composition; muscle mass; protein metabolism; enteral nutrition; ICU
MeSH Terms: conditions — Critical Illness; Muscle Weakness | interventions — beta-hydroxyisovaleric acid

STUDY DESIGN:
Intervention Model Description: Randomised, double blind, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation controlled by the Hospital Pharmacy Intervention product masked by the Hospital Pharmacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMB (beta-hydroxy beta-methylbutyrate) (Active Comparator): HMB, 1.5 g b.i.d., from day 4 to day 30 after ICU admission
  Interventions: Dietary Supplement: HMB (beta-hydroxy beta-methylbutyrate)
- Placebo (Placebo Comparator): Maltodextrin, 1.5 g b.i.d., from day 4 to day 30 after ICU admission
  Interventions: Dietary Supplement: HMB (beta-hydroxy beta-methylbutyrate)

INTERVENTIONS:
Dietary Supplement: HMB (beta-hydroxy beta-methylbutyrate) — 1.5 g, b.i.d., by the enteral route, from Day 4 to Day 30 (minimum 10 days)

SUMMARY:
The rapid decline of muscle mass and function in mechanically ventilated critically ill patients is associated with prolonged length of mechanical ventilation, prolonged intensive care (ICU) and hospital stay, increased ICU and hospital mortality, and prolonged impairment in physical function and quality of life. High protein feeding only partially attenuates the muscle loss. The aim is to study the impact of HMB (3 g/day) on the muscle mass of the critically ill patients from day 4 of their admission to maximum 30 days, but at least for 10 days.

DETAILED DESCRIPTION:
The rapid decline of muscle mass and function in mechanically ventilated critically ill patients is associated with poor outcome, and limitations of functional recovery. High protein feeding only partially attenuates the muscle loss. The aim is to study the impact of HMB (3 g/day) on the muscle mass of the critically ill patients from day 4 of their admission to maximum 30 days, but at least for 10 days. The study is testing a nutrition complement (HMB) that is included in feeding products registered for medical nutrition by Swiss Federal Authorities, but who do not provide sufficient protein quantities.

On days 4 and 15 after ICU admission, specific investigations will include: Ultrasound measurement of the muscle quadriceps femoris (CSA), bioimpedance analysis (BIA) of body composition, protein synthesis and catabolism using amino acid tracers. On D30 and D60: telephone contact to assess global health and mobility (SF-12).

ELIGIBILITY:
Inclusion Criteria:

* likely length of stay >5 days
* on mechanical ventilation
* likely survival >7 days
* full treatment
* functional gastro-intestinal tract
* presence of a central venous catheter

Exclusion Criteria:

* absence of consent
* less than 18 years patients
* gastro-intestinal dysfunction
* major burns >20% body surface
* admission for cardio-respiratory arrest or brain injury
* pregnancy or lactation
* diabetes mellitus (I and II)
* statin treatment
* patient on parenteral nutrition
* absence of central venous line
* participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Muscle mass of the thigh | Change between Day 4 and Day 15
  Ultrasound cross sectional area of the thigh, to quantify muscle loss

SECONDARY OUTCOMES:
Body composition | Change between Day 4 and Day 15
  Bioelectrical impedance analysis (BIA): calculation of body compartments, lean body mass, and phase angle
Protein synthesis and breakdown | Change between Day 4 and Day 15
  Multiple Amino acid tracer study: to detect chnges in protein metabolism between study start on day 4 and day 14 (i.e. after 10 days of intervention (HMB or placebo))
Muscle strength (global and handgrip) | Measurements on Days 4, 15, and 30
  Medical Research Council muscle score (MRC) to assess upper and lower limb strength, and handgrip strength (not always feasible in ICU patients) and determine magnitude of strength loss
Global Health and Mobility | on days 30 and 60
  Short Form 12 (SF-12) questionnaire to assess global health and mobility: range 12 to 56 points, the upper limit reflecting return to normal activity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne Hospitals, Lausanne, Switzerland

REFERENCES:
- [Result] Deutz NE, Matheson EM, Matarese LE, Luo M, Baggs GE, Nelson JL, Hegazi RA, Tappenden KA, Ziegler TR; NOURISH Study Group. Readmission and mortality in malnourished, older, hospitalized adults treated with a specialized oral nutritional supplement: A randomized clinical trial. Clin Nutr. 2016 Feb;35(1):18-26. doi: 10.1016/j.clnu.2015.12.010. Epub 2016 Jan 18. PMID 26797412
- [Result] Deutz NE, Pereira SL, Hays NP, Oliver JS, Edens NK, Evans CM, Wolfe RR. Effect of beta-hydroxy-beta-methylbutyrate (HMB) on lean body mass during 10 days of bed rest in older adults. Clin Nutr. 2013 Oct;32(5):704-12. doi: 10.1016/j.clnu.2013.02.011. Epub 2013 Mar 4. PMID 23514626
- [Result] Engelen MPKJ, Deutz NEP. Is beta-hydroxy beta-methylbutyrate an effective anabolic agent to improve outcome in older diseased populations? Curr Opin Clin Nutr Metab Care. 2018 May;21(3):207-213. doi: 10.1097/MCO.0000000000000459. PMID 29406417
- [Derived] Berger MM, Singer P, Wierzchowska-McNew RA, Viana MV, Ben-David IA, Pantet O, Perez C, Thaden JJ, Engelen MPKJ, Deutz NEP. Cytokine response to critical illness and its relation to amino acid metabolism. Clin Nutr. 2025 Sep;52:195-202. doi: 10.1016/j.clnu.2025.07.018. Epub 2025 Jul 26. PMID 40784156
- [Derived] Deutz NEP, Singer P, Wierzchowska-McNew RA, Viana MV, Ben-David IA, Pantet O, Thaden JJ, Ten Have GAM, Engelen MPKJ, Berger MM. Females have a different metabolic response to critical illness, measured by comprehensive amino acid flux analysis. Metabolism. 2023 May;142:155400. doi: 10.1016/j.metabol.2023.155400. Epub 2023 Jan 27. PMID 36717057
- [Derived] Pantet O, Viana MV, Engelen MPKJ, Deutz NEP, Gran S, Berger MM. Impact of ss-hydroxy-ss-methylbutyrate (HMB) in critically ill patients on the endocrine axis - A post-hoc cohort study of the HMB-ICU trial. Clin Nutr ESPEN. 2023 Feb;53:1-6. doi: 10.1016/j.clnesp.2022.11.017. Epub 2022 Nov 25. PMID 36657898
- [Derived] Viana MV, Becce F, Pantet O, Schmidt S, Bagnoud G, Thaden JJ, Ten Have GAM, Engelen MPKJ, Voidey A, Deutz NEP, Berger MM. Impact of beta-hydroxy-beta-methylbutyrate (HMB) on muscle loss and protein metabolism in critically ill patients: A RCT. Clin Nutr. 2021 Aug;40(8):4878-4887. doi: 10.1016/j.clnu.2021.07.018. Epub 2021 Jul 22. PMID 34358832
- [Derived] Deutz NEP, Singer P, Wierzchowska-McNew RA, Viana MV, Ben-David IA, Pantet O, Thaden JJ, Ten Have GAM, Engelen MPKJ, Berger MM. Comprehensive metabolic amino acid flux analysis in critically ill patients. Clin Nutr. 2021 May;40(5):2876-2897. doi: 10.1016/j.clnu.2021.03.015. Epub 2021 Mar 18. PMID 33946038